CLINICAL TRIAL: NCT06826352
Title: The Effects of Active and Passive Distraction Methods on Children's Pain, Fear and Anxiety During Invasive Procedures: a Randomized Controlled Clinical Trial
Brief Title: Effects of Active and Passive Distraction Methods on Children's Pain, Fear and Anxiety
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Gokoglu, Research assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/212
Record Dates: First submitted 2021-08-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pain; Fear; Anxiety
Keywords: pain; anxiety; fear; inpatient; child; video games; cartoons; clinical trial
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: The children assessed their own conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): There will be no intervention, just only an intravenous procedure will be applied by the nurse.
- Active Distraction (Experimental): The active distraction includes video games. In this group, children play video games during the procedure.
  Interventions: Behavioral: Active Distraction
- Passive Distraction (Experimental): Participation will be watch cartoon.
  Interventions: Behavioral: Passive Distraction

INTERVENTIONS:
Behavioral: Active Distraction — The video games will be played by children during the procedure.
  Arms: Active Distraction
Behavioral: Passive Distraction — The cartoons will be selected by the children related to their interests. The cartoons are included Pepee, Niloya, Tom and Jerry, Masha and The Bear and others.
  Arms: Passive Distraction

SUMMARY:
Background:

It is important that reduce children's pain, fear, and anxiety during the invasive procedures for building effective communication with children and their parents. Knowing the effective methods will be helpful to use in the pediatric clinical.

Objective:

This study aimed to determine the effects of watching cartoons, a passive distraction method and playing video games, an active distraction method, on the pain, fear and anxiety of 3- to 7-year-old children before, during and after invasive procedures.

Design:

A randomized controlled clinical trial

Setting(s):

General pediatric service of a training and research hospital in Istanbul

Participants:

The study sample included 105 children who were 3- to 7-years-old inpatients. The children were randomly assigned to the control (n=35), cartoon (n=35) and video game (n=35) groups.

Methods:

The data were collected using an introductory information form, the Oucher Pain Scale, the Children's State Anxiety Scale, and the Children's Fear Scale between November 26, 2019 and January 8, 2020. Data analysis was performed with SPSS software using the chi-squared test, and one-way and repeated measures ANOVA.

DETAILED DESCRIPTION:
The randomized controlled experimental study involved 105 children hospitalized in the general pediatric service from November 26, 2019, to January 8, 2020. All participants met the inclusion criteria and provided voluntary consent, along with their parents. The children will randomly be assigned to control and experimental groups using sealed envelopes, ensuring an unbiased selection process. Each of the three groups comprised 35 children: one control group receiving routine nursing practices and two experimental groups receiving routine nursing practices supplemented by either a passive distraction method (watching cartoons) or an active distraction method (playing video games). Data collection utilized several instruments, including The Information Form, The Oucher Pain Scale, The Children's State Anxiety Scale, and The Children's Fear Scale.

Before the data collection process:

The study's objectives will be thoroughly explained to the children and their parents in with written consent obtained from participations' parents. Those who consented will be randomly assigned to with another nurse. The children in the cartoon group chose a cartoon, while those in the video game group select a video game

Data Collection Tools included:

1. The Introductory Information Form: Comprising 12 questions regarding the patients' demographic information and the three scales utilized in the study.
2. The Oucher Pain Scale: Developed to assess children's pain levels, featuring six facial expressions that depict a spectrum of pain severity from "no pain" to "worst possible pain," providing a visual representation of pain.
3. The Children's State Anxiety Scale (CSAS): A visual scale designed for children aged 4 to 10, resembling a thermometer with a bulb at the bottom and ten horizontal lines. Children are instructed to indicate their level of anxiety or nervousness by placing a marker on the scale.
4. The Children's Fear Scale: This scale assesses children's fear levels through five facial expressions, ranging from a neutral face (0 = no anxiety) to a fearful face (4 = severe anxiety). It is primarily designed for children aged 5 to 10 but can be utilized for younger children with adequate language development.

Protocol:

There will be 3 groups. One of the groups will be a control group. The others are interventions group. One of intervention group is the passive distraction intervention which included watching cartoons. The other intervention group is the active distraction intervention which included playing video by mobile phone. During this method one of the nurses (not included the research) will be apply intravenous procedure.

Control Group: Children in the control group will be accompanied by a parent to the procedure room, where participants' vital signs will be recorded. Routine nursing practices, including bloodletting and intravenous procedure establishment, will be performed without any distraction methods. Pain, fear, and anxiety levels will be assessed by investigators two minutes before, during, and two minutes after the procedure.

Intervention Groups:

Passive Distractive Intervention Group Passive intervention group procedure is included cartoon watching. Children, in the Passive Distractive Intervention Group, will be accompanied by a parent to the procedure room, where participants' vital signs will be recorded. After that participations will be start watching cartoon, pain, fear, and anxiety levels will be measured at the same intervals as the control group, with observational recordings parameters made during the procedure. Parameters two minutes before, during, and two minutes after the procedure will be recorded by investigators to evaluate the overall impact of the distraction methods on pain, anxiety, and fear.

Cartoon Content: Prior to the procedure, children in the cartoon group select from a list of options, including Pepee, Niloya, Tom and Jerry, and Masha and The Bear. Cartoons time lapse is approximately 12 minutes. Participation begins to watch cartoon two minutes before the procedure and continued until its completion.

Active Distractive Intervention Group Children, in the Active Distractive Intervention Group, will be accompanied by a parent to the procedure room, where participants' vital signs will be recorded. Same procedure will be applied in this group. The participant will play the video with the hand he/she chooses to prevent the nurse's intravenous administration. Participants select the game, have no fixed time limits and continue until a play error occurred. Children can restart the game until the procedure concluded. Before the two minutes procedure the video will be started by participations and the parameters will be recorded two minutes before, during, and two minutes after the procedure by investigators Video Game Content: Children in the video game group were recommended games playable with one hand, such as Red Ball, Subway Surfers, Candy Crush Saga, and Wood Block Puzzle.

Children's pain, fear, and anxiety levels will be assessed using the Oucher Pain Scale, the Children's State Anxiety Scale, and the Children's Fear Scale before, during, and after the procedure. Vital signs, including pulse and oxygen saturation, will be measured using pulse oximetry, while blood pressure was assessed with a sphygmomanometer and stethoscope.

Study Hypotheses:

* Ho: The active and passive distraction methods have no effect on children's pain, fear, and anxiety.
* H1: The active and passive distraction methods effectively reduce children's pain during invasive procedures.
* H2: The active and passive distraction methods effectively reduce children's fear during invasive procedures.
* H3: The active and passive distraction methods effectively reduce children's anxiety during invasive procedures.
* H4: The active distraction method is more effective than the passive distraction method.

ELIGIBILITY:
Inclusion Criteria:

* between the ages 3-7 years
* first invasive procedures
* children do not have visual and auditory problems that prevent them from applying the scales
* developed the child's counting skills
* absence of developmental delay in language development
* absence of pain in the child before the procedure

Exclusion Criteria:

* second invasive procedures
* the parent didn't want to be voluntarily participate
* the child didn't want to be voluntarily participate

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
The Oucher Pain Scale | Pain score will be decrease during the procedure within the 3 minutues.
  Zero is equivalent to no pain and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
The Children's State Anxiety Scale | State Anxiety level will be decrease during the procedure within the 3 minutues.
  Zero is equivalent to no anxiety and 10 indicates the highest possible anxiety.

OTHER OUTCOMES:
The Children's Fear Scale | The fear will be decrease during the procedure within the 3 minutues.
  It has five facial expressions: a face with no expressions (0=no anxiety) to a face showing fear (4=severe anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Özge Sukut, PhD, Study Director — IUC
Locations (1):
- İstanbul University - Cerrahpasa, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ersig AL, Kleiber C, McCarthy AM, Hanrahan K. Validation of a clinically useful measure of children's state anxiety before medical procedures. J Spec Pediatr Nurs. 2013 Oct;18(4):311-9. doi: 10.1111/jspn.12042. Epub 2013 Jun 25. PMID 24094126
- [Background] Gerçeker GÖ, Ayar D, Özdemir Z, Bektaş M. Çocuk Anksiyete Skalası-Durumluluk ve Çocuk Korku Ölçeğinin Türk Diline Kazandırılması. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 2018; 11(1), 9-13.
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Beyer JE, Denyes MJ, Villarruel AM. The creation, validation, and continuing development of the Oucher: a measure of pain intensity in children. J Pediatr Nurs. 1992 Oct;7(5):335-46. PMID 1479552
- [Derived] Gokoglu A, Sukut O. Should I play or should I watch: the effects of active and passive distraction methods on children's pain, fear and anxiety during invasive procedures: a randomized controlled clinical trial. BMC Pediatr. 2025 Oct 28;25(1):875. doi: 10.1186/s12887-025-06188-1. PMID 41152799